CLINICAL TRIAL: NCT05604924
Title: A Clinical Trial to Evaluate Effectiveness of Virtual Reality Training Simulator for Cesarean Section
Brief Title: Virtual Reality Training Simulator for Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jee Yoon Park, Professor in osbtetrics, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B-2205-759-303
Record Dates: First submitted 2022-10-26; First posted 2022-11-03 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Virtual Reality
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants who received virtual reality training (Experimental)
  Interventions: Other: virtual reality training for cesarean section
- Participants who received similar contents in a standard PowerPoint presentation on a laptop (Placebo Comparator)
  Interventions: Other: virtual reality training for cesarean section

INTERVENTIONS:
Other: virtual reality training for cesarean section — Participants who received virtual reality training for cesarean section can learn the surgical procedures as if they were in a real field.

SUMMARY:
The goal of this is to determine the effectiveness of virtual reality training simulator for cesarean section.

Evaluate the effect of using VR surgery on the self-confidence and knowledge of cesarean section procedures.

DETAILED DESCRIPTION:
A single center randomized controlled trial (RCT) was performed. The participants were obstetrics residents, fellows and residents in other majors with limited experience in performing cesarean section. The primary outcome measures were the self-assessment scores of trainee confidence using a virtual reality training and an objective assessment of the cognitive skills. The participants were randomly divided into a study group of VR training group and a control group. Participants in the study group used the VR application. The control group participants used similar content in a standard PowerPoint presentation on a laptop.

ELIGIBILITY:
Inclusion Criteria:

* Residents and fellows receiving training at Seoul National University Bundang Hospital and who wish to participate in this study

Exclusion Criteria:

* If trainee refuse to participate in this study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
improvement on the knowledge of cesarean section procedures. | 1 month after examination
  After using VR training, the test scores cesarean section procedures.
improvement on the self-confidence of cesarean section procedures. | 1 month after examination
  After using VR training, the self-assessment scores of trainee confidence via questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeong-gi Do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided